CLINICAL TRIAL: NCT00442416
Title: A Two-arm, Randomized, Open-label, Multicenter Study of Safety and Efficacy of Monthly Injections of RO0503821 Versus Epoetin Alfa in Peritoneal Dialysis Patients Who Self Inject or Receive In-center Injections.
Brief Title: A Study of Subcutaneous Mircera for the Treatment of Anemia in Peritoneal Dialysis Patients.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic decision unrelated to safety or efficacy
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20338
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-07

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa; continuous erythropoietin receptor activator

ARMS (2):
- RO0503821 (Experimental): Eligible participants will be administered RO0503821 (methoxy polyethylene glycol-epoetin beta [Mircera]) subcutaneously (SC) every month for eight months (6 months of titration period [TP] and two months of evaluation period [EP] and 15-days following the final study visit (9 months post randomization). The first dose of Mircera (120, 200, or 360 mcg) will be based upon the dose of epoetin alfa received 1 to 2 weeks prior to administration of study drug, while subsequent doses will be adjusted to maintain haemoglobin (Hb) concentrations within target of >=10.0 gram per decilitre (g/dL) and <=12.0 g/dL. Participants who self-administered/visited to clinics for erythropoiesis stimulating agent (ESA) dosing prior to randomization will continue to do so.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Epoetin Alfa (Active Comparator): Eligible participants will be administered epoetin alfa SC as per the standard of care for eight months (TP and EP), and will be followed-up for 15 days following the final study visit. Participants who self-administered/visited to clinics for ESA dosing prior to randomization will continue to do so.
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: Epoetin alfa — As prescribed, SC
  Arms: Epoetin Alfa
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 120-360 micrograms SC monthly, starting dose
  Arms: RO0503821

SUMMARY:
This 2 arm study will compare the efficacy of monthly Mircera and epoetin alfa in peritoneal dialysis patients who self-inject at home or receive in-centre injections. The safety of subcutaneous (sc) Mircera and injection site reactions and patient satisfaction will also be assessed. Eligible patients will be randomized either to receive monthly sc injections of Mircera (and will be switched from sc epoetin alfa) at a starting dose of 120-360 micrograms, or to remain on standard of care sc epoetin alfa. Dose adjustments will be permitted to reach/maintain a hemoglobin level of 10-12g/dL. The anticipated time on study treatment is 3-12 months, and the target sample size is 380 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic kidney disease stage V;
* on peritoneal dialysis for 3 months prior to screening;
* on epoetin alfa sc >=3 months prior to screening.

Exclusion Criteria:

* patients expecting to change dialysis modality over course of study;
* patients hospitalized during previous 3 months for any clinically significant condition;
* active malignancy;
* bleeding episode necessitating transfusion, or overt gastrointestinal bleeding within 3 months prior to screening;
* transfusion of red blood cells within 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (29):
- United States (29):
  - Birmingham, Alabama
  - Bakersfield, California
  - Chula Vista, California
  - Mountain View, California
  - San Leandro, California
  - Simi Valley, California
  - Whittier, California
  - Lakewood, Colorado
  - Stamford, Connecticut
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Augusta, Georgia
  - Marietta, Georgia
  - Wichita, Kansas
  - Detroit, Michigan
  - Pontiac, Michigan
  - Flushing, New York
  - Syracuse, New York
  - Williamsville, New York
  - Dayton, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Lewistown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Dyersburg, Tennessee
  - San Antonio, Texas
  - Tyler, Texas
  - Alexandria, Virginia
  - Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the United States from 27 February 2007 to 01 January 2008. The study was prematurely terminated during enrolment due to legal reasons.
Pre-assignment Details: A total of 80 participants were randomized, of which 78 participants received the study drug and 2 participants did not receive the study drug nor had post baseline safety assessments.
Groups:
- RO0503821: Eligible participants were administered RO0503821 (methoxy polyethylene glycol-epoetin beta [Mircera]) subcutaneously (SC) every month for eight months (6 months of titration period [TP] and two months of evaluation period [EP] and 15-days following the final study visit (9 months post randomization). The first dose of Mircera (120, 200, or 360 mcg) was based upon the dose of epoetin alfa received 1 to 2 weeks prior to administration of study drug, while subsequent doses were adjusted to maintain haemoglobin (Hb) concentrations within target of >=10.0 gram per decilitre (g/dL) and <=12.0 g/dL. Participants who self-administered/visited to clinics for erythropoiesis stimulating agent (ESA) dosing prior to randomization continued to do so.
- Epoetin Alfa: Eligible participants were administered epoetin alfa SC as per the standard of care for eight months (TP and EP), and were followed-up for 15 days following the final study visit. Participants who self-administered/visited to clinics for ESA dosing prior to randomization continued to do so.
Period: Overall Study
Arm/Group | RO0503821 | Epoetin Alfa
Started | 39 | 41
Completed | 2 | 2
Not Completed | 37 | 39
Not completed — Adverse Event | 4 | 1
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrew consent | 1 | 2
Not completed — Administrative/Other | 27 | 33

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of the study drug and had at least one post-baseline safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | RO0503821 | Epoetin Alfa | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (12.59) | 53.6 (15.86) | 56.0 (14.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hb Concentration to Average Over the Evaluation Period
Description: Mean change in Hb concentration from Baseline (Day [D] 0) to average during the evaluation period (Month 7 to 9) is reported.
Time Frame: From Baseline (D 0) to 9 months
Population: Per-protocol population included all randomized participants who received at least one dose of the study drug and met all study entry criteria with no major protocol violations. Participants with available data at the time of evaluation were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 33 | 35
g/dL | -0.32 (1.31) | 0.51 (1.33)

2. Secondary Outcome: Percentage of Participants With Safety-Related Hb Measures
Description: Safety-related Hb measures included percentage of participants with Hb value > 13 g/dL, 13.5 g/dL, increase in Hb value from baseline by > 2 g/dL or decrease in Hb value from baseline by > 2 g/dL at any time during the study.
Time Frame: Up to Month 9
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
Percentage of participants
  Hb value > 13 g/dL | 34 | 33
  Hb value > 13.5 g/dL | 13 | 13
  Increase in Hb value > 2 g/dL | 24 | 20
  Decrease in Hb value > 2 g/dL | 16 | 5

3. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Participants with marked laboratory abnormalities in hematology and clinical chemistry parameters are reported. Hematology laboratory parameters included hematocrit fraction, hemoglobin, platelets, white blood cells (WBCs) and clinical chemistry parameters included aspartate aminotransferase ([AST], alanine aminotransferase ([ALT], creatine phosphokinase (CPK), alkaline phosphatase, albumin, potassium, fasting glucose and phosphate.
Time Frame: Up to Month 9
Population: Safety population included all participants who received at least one dose of the study drug and had at least one post-baseline safety assessment. Participants with available data at the time of evaluation were denoted as 'n'.
Measure: Number; unit: Participants
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
Participants
  Hematocrit - Low (n = 38, 40) | 8 | 3
  Hemoglobin - Low (n = 38, 40) | 11 | 3
  Platelets - High (n = 38, 40) | 0 | 1
  Platelets - Low (n = 38, 40) | 1 | 0
  WBCs - Low (n = 38, 40) | 0 | 1
  AST - High (n = 37, 40) | 0 | 2
  ALT - High (n = 38, 40) | 1 | 2
  CPK- High (n = 37, 40) | 7 | 3
  Alkaline phosphatase - High, (n = 37, 40) | 1 | 1
  Albumin - Low (n = 38, 40) | 6 | 0
  Potassium - High (n = 38, 40) | 3 | 4
  Fasting glucose - High (n = 38, 40) | 6 | 5
  Fasting glucose - Low (n = 38, 40) | 0 | 1
  Phosphate - High (n = 38, 40) | 17 | 7

4. Secondary Outcome: Mean Change From Baseline in Iron
Description: Adequate iron status is prerequisite to achieve and maintain target Hb levels. Mean change from Baseline (D 0) in iron to D1 of Months 2, 3, 4, 5, 6, 7, 8 is reported.
Time Frame: From Baseline (D 0) to Month (M) 2, M3, M4, M5, M6, M7, M8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micromole per litre
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
micromole per litre
  M2 (n = 33, 31) | 3.4 (7.25) | 1.8 (5.07)
  M3 (n = 29, 29) | 3.9 (5.39) | -1.3 (5.87)
  M4 ( n = 22,24) | 2.0 (6.97) | 0.2 (3.26)
  M5 (n = 18, 17) | 3.1 (7.66) | 0.9 (2.54)
  M6 (n = 13, 10) | 2.9 (8.33) | 0.6 (3.94)
  M7 (n = 8, 6) | 3.4 (5.94) | -1.3 (4.84)
  M8 (n = 2, 3) | 11.0 (13.80) | 7.7 (13.80)

5. Secondary Outcome: Mean Change From Baseline in Ferritin
Description: Adequate iron status is prerequisite to achieve and maintain target Hb levels. Mean change from Baseline (D 0) in ferritin to D1 of M2, 3, 4, 5, 6, 7, and 8 is reported.
Time Frame: From Baseline (D 0) to M2, M3, M4, M5, M6, M7, M8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microgram per litre
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
microgram per litre
  M2 (n = 32, 29) | 59 (128.8) | -1 (129.5)
  M3 (n = 28, 27) | 83 (195.1) | -37 (114.2)
  M4 ( n = 21,22) | 48 (319.7) | -24 (155.4)
  M5 (n = 17, 16) | 85 (242.0) | -70 (149.6)
  M6 (n = 12, 9) | 86 (226.1) | -105 (187.8)
  M7 (n = 7, 6) | 55 (117.1) | -120 (166.3)
  M8 (n = 2, 3) | -59 (176.8) | -99 (36.8)

6. Secondary Outcome: Mean Change From Baseline in Transferrin Saturation
Description: Adequate iron status is prerequisite to achieve and maintain target Hb levels. Mean change from Baseline (D 0) in transferrin to D1 of M2, 3, 4, 5, 6, 7, and 8 is reported.
Time Frame: From Baseline (D 0) to M2, M3, M4, M5, M6, M7, M8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Transferrin Saturation
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
Percentage of Transferrin Saturation
  M2 (n = 33, 31) | 7.10 (15.32) | 4.08 (10.39)
  M3 (n = 29, 29) | 8.51 (12.04) | -2.44 (13.33)
  M4 ( n = 22,24) | 4.55 (17.08) | 1.36 (8.52)
  M5 (n = 18, 17) | 5.94 (16.21) | 3.47 (6.91)
  M6 (n = 13, 10) | 7.07 (18.10) | 0.39 (10.79)
  M7 (n = 8, 6) | 8.59 (12.20) | -1.80 (10.90)
  M8 (n = 2, 3) | 24.13 (27.83) | 15.13 (23.28)

7. Secondary Outcome: Mean Change From Baseline in Serum Transferrin
Description: Adequate iron status is prerequisite to achieve and maintain target Hb levels. Mean change from Baseline (D 0) in serum transferrin to D1 of M2, 3, 4, 5, 6, 7, and 8 is reported.
Time Frame: From Baseline (D 0) to M2, M3, M4, M5, M6, M7, M8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram (mg) per dL
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
milligram (mg) per dL
  M2 (n = 15, 14) | -9.27 (20.38) | -5.00 (16.06)
  M3 (n = 12,15) | -0.25 (24.68) | -7.73 (19.56)
  M4 ( n = 8, 14) | 7.25 (16.02) | -4.21 (20.75)
  M5 (n = 9, 11) | 9.89 (29.36) | -6.64 (23.68)
  M6 (n = 6, 6) | 10.50 (27.19) | 1.50 (16.84)
  M7 (n = 4, 5) | 2.50 (24.06) | -5.60 (24.30)
  M8 (n = 2, 2) | -15.50 (9.19) | -6.50 (12.02)

8. Secondary Outcome: Mean Change From Baseline in Total Iron-binding Capacity
Description: Adequate iron status is prerequisite to achieve and maintain target Hb levels. Mean change from Baseline (D 0) in total Iron-binding Capacity to D1 of M2, 3, 4, 5, 6, 7, and 8 is reported.
Time Frame: From Baseline (D 0) to M2, M3, M4, M5, M6, M7, M8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg per dL
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
mg per dL
  M2 (n = 18, 17) | 20.94 (67.80) | 1.94 (29.47)
  M3 (n = 17,14) | -3.29 (45.64) | -9.57 (25.58)
  M4 ( n = 12, 9) | 15.17 (41.51) | 4.67 (19.25)
  M5 (n = 9, 5) | 19.67 (53.53) | 8.60 (7.89)
  M6 (n = 7, 4) | 9.29 (62.96) | 21.25 (48.34)
  M7 (n = 4, 1) | 3.25 (85.99) | 3.00 (NA) — Data was available for only one participant; therefore, standard deviation cannot be calculated.
  M8 (n = 0, 1) | NA (NA) — Data was not recorded at this visit. | -43.00 (NA) — Data was available for only one participant; therefore, standard deviation cannot be calculated.

9. Secondary Outcome: Mean Change From Baseline in Temperature
Time Frame: From Baseline (D 0) to D1 and D15 of M7, M8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
Degree Celsius
  M7 D1 (n = 9, 6) | -0.0 (0.43) | -0.3 (1.03)
  M7 D15 (n = 5, 3) | 0.2 (0.54) | -0.7 (1.44)
  M8 D1 (n = 2, 3) | 0.5 (0.14) | -0.5 (0.95)
  M8 D15 (n = 2, 2) | 0.1 (0.21) | -0.4 (0.07)

10. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure
Time Frame: From Baseline (D 0) to D1 and D15 of M7, M8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
millimeter of mercury
  SBP at M7 D1 (n = 9, 6) | 3 (18.4) | 9 (22.7)
  DBP at M7 D1 (n = 9, 6) | 3 (10.2) | 2 (6.9)
  SBP at M7 D15 (n = 5, 3) | 5 (13.3) | -7 (14.2)
  DBP at M7 D15 (n = 5, 3) | 1 (10.7) | -2 (2.5)
  SBP at M8 D1 (n = 2, 3) | 7 (12.7) | 5 (19.3)
  DBP at M8 D1 (n = 2, 3) | -5 (2.1) | -1 (7.9)
  SBP at M8 D15 (n = 2, 2) | 6 (2.8) | -6 (26.9)
  DBP at M8 D15 (n = 2, 2) | -6 (10.6) | -5 (10.6)

11. Secondary Outcome: Mean Change From Baseline in Pulse Rate
Time Frame: From Baseline (D 0) to D1 and D15 of M7, M8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
Beats per minute
  M7 D1 (n = 9, 6) | -2 (11.0) | -2 (10.6)
  M7 D15 (n = 5, 3) | 1 (13.3) | 3 (3.1)
  M8 D1 (n = 2, 3) | -7 (0.0) | 2 (4.4)
  M8 D15 (n = 2, 2) | -4 (3.5) | 7 (6.4)

12. Secondary Outcome: Mean Change From Baseline in Weight
Time Frame: From Baseline (D 0) to D1 and D15 of M7, M8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
kilogram
  M7 D1 (n = 9, 6) | 0.5 (3.56) | 3.2 (3.46)
  M7 D15 (n = 5, 3) | 1.2 (2.93) | 1.1 (2.14)
  M8 D1 (n = 2, 3) | 3.0 (4.74) | 1.9 (1.57)
  M8 D15 (n = 2, 2) | 1.5 (3.04) | 2.5 (2.33)

13. Secondary Outcome: Number of Participants With Anti-erythropoietin Antibody in Human Serum
Description: Erythropoietin is human protein which helps to make more RBCs and is used for the treatment of anemia of chronic kidney disease. However, during treatment with erythropoietin, anti-erythropoietin antibody (Anti-EPO) may develop in human serum. These antibodies have been shown to cross-react with all ESAs and leads to failure to respond to treatment. Number of participants with anti-EPO antibody that are quantifiable and those that were "below the limit of quantification (BLQ)" at Baseline (Day 0) and Visit 17 (Month 9 [M 9]) or final visit/early termination in human serum samples are reported.
Time Frame: Up to Month 9
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
Participants
  Quantifiable at Baseline | 2 | 1
  BLQ at Baseline | 33 | 37
  Quantifiable at M 9 final visit/early termination | 1 | 4
  BLQ at M 9 final visit/early termination | 29 | 34

14. Secondary Outcome: Number of Participants With Anti-RO0503821 Antibody in Human Serum
Description: RO0503821 is a chemically modified erythropoietin which helps to make more RBCs and is used for the treatment of anemia of chronic kidney disease. However, during treatment with RO0503821, anti-RO0503821 antibody may develop in human serum. These antibodies have been shown to cross-react with all ESAs and leads to failure to respond. Number of participants with anti- RO0503821 antibody that are quantifiable and those that were "BLQ" at Baseline (Day 0) and Visit 17 (M 9) or final visit/early termination in human serum samples are reported.
Time Frame: Up to Month 9
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | RO0503821
Number analyzed (Participants) | 36
Participants
  Quantifiable at Baseline | 0
  BLQ at Baseline | 35
  Quantifiable at M 9 final visit/early termination | 0
  BLQ at M 9 final visit/early termination | 29

15. Secondary Outcome: Number of Participants With Any AEs, Any Serious Adverse Events and Death
Description: An AE is untoward medical occurrence in a participant who received the study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is with any of the following outcomes: Death, initial or prolonged inpatient hospitalisation, life-threatening experience, persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 9 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | RO0503821 | Epoetin Alfa
Number analyzed (Participants) | 38 | 40
Participants
  Any AEs | 24 | 23
  Any SAEs | 11 | 2
  Death | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 9 months
Description: Safety population included all participants who received at least one dose of the study drug and had at least one post-baseline safety assessment.
Arm/Group | RO0503821 | Epoetin Alfa
Serious Adverse Events (participants affected / at risk) | 11/38 | 2/40
Other Adverse Events (participants affected / at risk) | 18/38 | 15/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (N=38) | Epoetin Alfa (N=40)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (N=38) | Epoetin Alfa (N=40)
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Peritonitis (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 2 | 0 — General disorders and administration site conditions
Fatigue (General disorders) | 5 | 0 — General disorders and administration site conditions
Bronchitis (Infections and infestations) | 2 | 1
Catheter site infection (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 2
Postoperative wound infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypertension (Vascular disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The study was prematurely terminated during enrollment period due to legal reasons. Therefore, the planned statistical analysis of the primary endpoint was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.